CLINICAL TRIAL: NCT07286370
Title: A Phase 2a, Observer-Blind, Randomized, Controlled, Age-De-Escalation, Single-center Interventional Study to Evaluate the Safety, Reactogenicity, and Immune Response of the GVGH iNTS-TCV Vaccine Against Invasive Nontyphoidal Salmonella (iNTS) Disease and Typhoid Fever, Including Dose and Schedule Finding in Infants, in Africa
Brief Title: A Study to Evaluate Safety, Reactogenicity, and Immune Response of GVGH iNTS-TCV Vaccine Against Invasive Nontyphoidal Salmonella Disease and Typhoid Fever in Infants
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 223550
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Salmonella Infections
Keywords: Salmonella-typhoid conjugate (iNTS-TCV) vaccine; Typhoid fever; Infants; Safety; Reactogenicity; Immunogenicity
MeSH Terms: conditions — Salmonella Infections; Typhoid Fever | interventions — 13-valent pneumococcal vaccine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Data will be collected in an observer-blind manner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Step 1a- Group 1 iNTS-TCV low dose (6 MOA) (Experimental): Participants 6 MOA receive 3 doses of a low dose of iNTS-TCV at Day 1, Day 85 and Day 337.
  Interventions: Biological: Low dose of iNTS-TCV
- Step 1a Group 2- Control group (6MOA) (Active Comparator): Participants 6 MOA receive TYPHIBEV at Day 1, pneumococcal polysaccharide conjugate vaccine (13 valent) (Prevenar 13) at Day 85, and Nimenrix at Day 337.
  Interventions: Biological: TYPHIBEV; Combination Product: Prevenar 13; Combination Product: Nimenrix
- Step 1b Group 3- iNTS-TCV full dose (6 MOA) (Experimental): Participants 6 MOA receive 3 doses of a full dose of iNTS-TCV at Day 1, Day 85 and Day 337.
  Interventions: Biological: Full dose of iNTS-TCV
- Step 1b Group 4- iNTS-TCV full dose + Prevenar 13 (6 MOA) (Experimental): Participants 6 MOA receive 2 doses of a full dose of iNTS-TCV at Day 1 and Day 337 and 1 dose of Prevenar 13 at Day 85.
  Interventions: Biological: Full dose of iNTS-TCV; Combination Product: Prevenar 13
- Step 1b Group 5- Control Group (6 MOA) (Active Comparator): Participants 6 MOA receive TYPHIBEV at Day 1, Prevenar 13 at Day 85, and Nimenrix at Day 337.
  Interventions: Biological: TYPHIBEV; Combination Product: Prevenar 13; Combination Product: Nimenrix
- Step 1c- Group 6- iNTS-TCV low dose (6 WOA) (Experimental): Participants 6 WOA receive 3 doses of a low dose of iNTS-TCV at Day 1, Day 57 and Day 232.
  Interventions: Biological: Low dose of iNTS-TCV
- Step 1c- Group 7- Control Group (6 WOA) (Active Comparator): Participants 6 WOA receive 2 doses of Nimenrix at Day 1 and Day 57, and 1 dose of TYPHIBEV at Day 232
  Interventions: Biological: TYPHIBEV; Combination Product: Nimenrix
- Step 1d- Group 8- iNTS-TCV full dose (6 WOA) (Experimental): Participants 6 WOA receive 3 doses of a full dose of iNTS-TCV at Day 1, Day 57 and Day 232.
  Interventions: Biological: Full dose of iNTS-TCV
- Step 1d- Group 9- Control Group (6 WOA) (Active Comparator): Participants 6 WOA receive 2 doses of Nimenrix at Day 1 and Day 57, and 1 dose of TYPHIBEV at Day 232
  Interventions: Biological: TYPHIBEV; Combination Product: Nimenrix
- Step 2- Group 10- iNTS-TCV low dose (6 WOA) (Experimental): Participants 6 WOA receive 3 doses of a low dose of iNTS-TCV at Day 1, Day 57 and Day 232.
  Interventions: Biological: Low dose of iNTS-TCV
- Step 2- Group 11- iNTS-TCV low dose+ Saline Group (6 WOA) (Experimental): Participants 6 WOA receive 1 dose of a saline on Day 1 and 2 doses of low dose of iNTS-TCV at Day 57 and Day 232.
  Interventions: Biological: Low dose of iNTS-TCV; Drug: Saline
- Step 2- Group 12- iNTS-TCV full dose (6 WOA) (Experimental): Participants 6 WOA receive 3 doses of a full dose of iNTS-TCV at Day 1, Day 57 and Day 232.
  Interventions: Biological: Full dose of iNTS-TCV
- Step 2- Group 13- iNTS-TCV full dose+ Saline Group (6 WOA) (Experimental): Participants 6 WOA receive 1 dose of saline on Day 1 and 2 doses of full dose of iNTS-TCV at Day 57 and Day 232.
  Interventions: Biological: Full dose of iNTS-TCV; Drug: Saline
- Step 2- Group 14 - Control Group (6 WOA) (Active Comparator): Participants 6 WOA receive 2 doses of Nimenrix at Day 1 and Day 57, and 1 dose of TYPHIBEV at Day 232
  Interventions: Biological: TYPHIBEV; Combination Product: Nimenrix

INTERVENTIONS:
Biological: Low dose of iNTS-TCV — Low dose of iNTS-TCV vaccine will be administered.
  Arms: Step 1a- Group 1 iNTS-TCV low dose (6 MOA); Step 1c- Group 6- iNTS-TCV low dose (6 WOA); Step 2- Group 10- iNTS-TCV low dose (6 WOA); Step 2- Group 11- iNTS-TCV low dose+ Saline Group (6 WOA)
Biological: Full dose of iNTS-TCV — Full dose of iNTS-TCV vaccine will be administered.
  Arms: Step 1b Group 3- iNTS-TCV full dose (6 MOA); Step 1b Group 4- iNTS-TCV full dose + Prevenar 13 (6 MOA); Step 1d- Group 8- iNTS-TCV full dose (6 WOA); Step 2- Group 12- iNTS-TCV full dose (6 WOA); Step 2- Group 13- iNTS-TCV full dose+ Saline Group (6 WOA)
Biological: TYPHIBEV — TYPHIBEV vaccine will be administered.
  Other Names: Typhoid Vi-CRM197 conjugate vaccine
  Arms: Step 1a Group 2- Control group (6MOA); Step 1b Group 5- Control Group (6 MOA); Step 1c- Group 7- Control Group (6 WOA); Step 1d- Group 9- Control Group (6 WOA); Step 2- Group 14 - Control Group (6 WOA)
Combination Product: Prevenar 13 — Prevenar 13 vaccine will be administered.
  Arms: Step 1a Group 2- Control group (6MOA); Step 1b Group 4- iNTS-TCV full dose + Prevenar 13 (6 MOA); Step 1b Group 5- Control Group (6 MOA)
Combination Product: Nimenrix — Nimenrix vaccine will be administered.
  Other Names: meningococcal groups A, C, W-135 and Y conjugate vaccine
  Arms: Step 1a Group 2- Control group (6MOA); Step 1b Group 5- Control Group (6 MOA); Step 1c- Group 7- Control Group (6 WOA); Step 1d- Group 9- Control Group (6 WOA); Step 2- Group 14 - Control Group (6 WOA)
Drug: Saline — Saline will be administered.
  Arms: Step 2- Group 11- iNTS-TCV low dose+ Saline Group (6 WOA); Step 2- Group 13- iNTS-TCV full dose+ Saline Group (6 WOA)

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity, and immune response induced by the GlaxoSmithKline Biologicals SA (GSK) Vaccines Institute for Global Health (GVGH) invasive nontyphoidal Salmonella-typhoid conjugate (iNTS-TCV) vaccine in infants with the first dose administered at 6 months of age (MOA) or 6 weeks of age (WOA).

ELIGIBILITY:
Inclusion Criteria:

Participants must:

1. Have signed/thumb-printed, voluntary, informed consent provided for them by their parent/Legally Authorized Representative (LAR) prior to performance of any study-specific procedure.
2. Be a male or female infant aged 6 months (±2 weeks) or 6 weeks (+2 weeks) of age at the time of the first study vaccination.
3. Have a parent/LAR, who can and will comply with the requirements of the protocol.
4. Healthy as established by medical history, clinical examination, and laboratory assessment.
5. Have received all routine childhood vaccinations as per the age.
6. Have been born at full term (>=37 weeks gestation) based on maternal report and additional antenatal records if available.
7. Have a parent/LAR who is willing to avoid the administration of local herbal/traditional medications (including topical treatments) throughout the study period and who is willing to consult, as applicable, the study team prior to the use on other medications including over the-counter medications not supplied by the study team (except in the case of an emergency) throughout the study period.
8. Have a readily identifiable place of residence within a reasonable travelling distance of the study site.
9. Have a parent/LAR with a means of telephone contact.
10. Have a parent/LAR who is willing to avoid vaccinations not provided by the study team throughout the participant's enrollment in the study. All routine Essential Programme on Immunization (EPI) vaccines due during the study (outside those given concurrently with the study vaccines/controls) will also be administered by the study team.

Exclusion Criteria:

Participants must not:

1. Have had a known infection with STm, SEn or S. Typhi.
2. Have a history of allergic reactions to any prior vaccination or components of the investigational or control vaccines.
3. Hypersensitivity to latex.
4. History of any reaction or hypersensitivity likely to be exacerbated by any component of the study interventions.
5. Have any history of anaphylaxis or other life-threatening allergic reactions.
6. Have any confirmed or suspected congenital or acquired immunosuppressive or immunodeficient condition, based on medical history and physical examination.
7. Have any acute or chronic, clinically significant pulmonary, cardiovascular, hepatobiliary, gastrointestinal, renal, neurological, or hematological abnormality or illness, as determined by medical history, physical examination, and (when applicable) baseline laboratory assessments. Known sickle cells disease (but not sickle cell trait) is an exclusion.
8. Have a bleeding or coagulation disorder contraindicating intramuscular injections or any other condition that in the judgment of the Investigator would make intramuscular injection unsafe.
9. Have a documented fever (axillary temperature ≥37.5ºC) at the time of enrollment/dosing or within the 48 hours preceding dosing (temporary exclusion if remains age-eligible/within the allowed interval of dosing).
10. Have clinically significant (moderate in severity) acute illness on the day of vaccination (temporary exclusion if remains age-eligible within the allowed dosing window).
11. Have any screening/last pre-dosing safety laboratory test (if applicable) with a toxicity score of ≥3 or a value judged to be clinically significant by the study clinician.
12. Have HIV, hepatitis B, or hepatitis C based on baseline serological assessment (these serological evaluations are only required during the screening phase).
13. Be known to have been vertically exposed to HIV based on maternal history and baseline serological assessment in the participant (maternal screening for HIV will not be undertaken).
14. Have a positive rapid diagnostic test (RDT) (or blood film) for malaria (temporary exclusion if remains age-eligible).
15. Have major congenital defects, as assessed by the Investigator.
16. Recurrent history or uncontrolled neurological disorders or any neuroinflammatory (including, but not limited to demyelinating disorders, encephalitis or myelitis of any origin), congenital neurological conditions, encephalopathies, or any history of seizures.
17. Be malnourished at Screening Visit, defined as WHO weight for length Z-score less than -2 standard deviation (SD).
18. Any other clinical condition that might pose additional risk to the participant as a result of participation in the clinical study.
19. Have used traditional or local herbal medications, including topical medications, in the 14 days prior to enrollment
20. Have a history of chronic administration of immune-modifying drugs (defined as more than 14 consecutive days) and/or planned use of long-acting immune-modifying treatments at any time up to the end of the study.

    1. for corticosteroids, this will mean prednisone equivalent >=0.5mg/kg/day with maximum of 20 mg/day for pediatric participants). The use of inhaled/per nasal and topical steroids are allowed.
    2. long-acting immune-modifying drugs including among others immunotherapy (eg, TNF-inhibitors), monoclonal antibodies, antitumoral medication.
21. Prior receipt of a typhoid vaccine, or an experimental iNTS or GMMA vaccine.
22. Use of any investigational or non-registered product (drug, vaccine, or medical device) other than the study intervention during the period starting 28 days before the first dose of study intervention (Day -28 to Day 1), or planned use during the study period.
23. A vaccine not foreseen by the study protocol administered during the period starting at 14 days before the first dose and ending 14 days after the last dose of study interventions administration for live vaccines or 7 days in case of inactivated vaccines, with the exception of flu vaccines or Coronavirus disease 2019 (COVID-19) vaccine which may be considered on a case-by-case basis.
24. Have been administered immunoglobulins and/or any blood products or plasma derivatives, or bone marrow transplantation, during the period starting 3 months before the first dose of study interventions or planned administration during the study period.
25. Concurrently participating in another interventional clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non investigational intervention (drug or invasive medical device).
26. Have any other factor which, in the opinion of the Investigator, might pose additional risk to the participant or substantially compromise data quality or the evaluation of study endpoints.
27. Any study personnel or their immediate dependents, family, or household members.
28. Have plans to travel outside the study area for an extended duration during the period of study participation.
29. Child in care.

Ages: 6 Weeks to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 537 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2028-04-27 (Estimated); Study Completion 2028-04-27 (Estimated)

PRIMARY OUTCOMES:
Number of participants with solicited administration site events during 7 days after each study intervention administration [for infants 6 MOA] | At Day 1, Day 85 and Day 337
  Solicited administration site events included pain, redness, and swelling.
Number of participants with solicited systemic events during 7 days after each study intervention administration [for infants 6 MOA] | At Day 1, Day 85 and Day 337
  Solicited systemic events included Fever, Irritability/Fussiness, Loss of appetite, Somnolence (sleepiness/drowsiness) and Vomiting. Fever is defined as body temperature more than or equal to (>=) 37.5 degrees Celsius (°C), measured from axilla.
Number of participants with unsolicited adverse events (AEs) during 28 days after each study intervention administration [for infants 6 MOA] | At Day 1, Day 85 and Day 337
  An unsolicited AE is defined as an AE that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events.
Number of participants with serious adverse events (SAEs) [for infants 6 MOA] | From the first study intervention administration (Day 1) until study end (Day 505).
  An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, results in abnormal pregnancy outcomes or any other situation based on appropriate medical or scientific judgement.
Number of participants with AEs/SAEs leading to withdrawal from the study or discontinuation of study intervention [for infants 6 MOA] | From the first study intervention administration (Day 1) until study end (Day 505).
Number of participants with laboratory abnormalities [for infants 6 MOA] | At 7 days after each study intervention administration (Day 8, Day 92 and Day 344).
Number of participants with solicited administration site events during 7 days after each study intervention administration [for infants 6 WOA] | At Day 1, Day 57 and Day 232
Number of participants with solicited systemic events during 7 days after each study intervention administration [for infants 6 WOA] | At Day 1, Day 57 and Day 232
Number of participants with unsolicited adverse events (AEs) during 28 days after each study intervention administration [for infants 6 WOA] | At Day 1, Day 57 and Day 232
Number of participants with SAEs [for infants 6 WOA] | From the first study intervention administration (Day 1) until study end (Day 400).
Number of participants with AEs/SAEs leading to withdrawal from the study or discontinuation of study intervention [for infants 6 WOA] | From the first study intervention administration (Day 1) until study end (Day 400).
Number of participants with laboratory abnormalities [for infants 6 WOA] | At 7 days after each study intervention administration (Day 8, Day 64 and Day 239).
Geometric Mean concentration (GMC) ratio of anti- S. typhimurium (STm) and anti- Salmonella Enteritidis (SEn) O-antigen (OAg) immunoglobulin G (IgG) [for infants 6 MOA] | At 28 days after the second study intervention administration (Day 113)
GMC ratio of anti-Vi IgG [for infants 6 MOA] | At 28 days after the first study intervention administration (Day 29)
GMC ratio of anti-STm and anti-SEn OAg IgG concentrations [for infants 6 WOA] | At 28 days after the third study intervention administration (Day 260)
GMC ratio of anti-Vi IgG [for infants 6 WOA] | At 28 days after the third study intervention administration (Day 260)

SECONDARY OUTCOMES:
GMC of anti-STm OAg, anti-SEn OAg and anti-Vi IgG before each study intervention administration [for infants 6 MOA] | At Day 1, Day 85 and Day 337
GMC of anti-STm OAg, anti-SEn OAg and anti-Vi IgG 28 days after each study intervention administration [for infants 6 MOA] | At Day 29, Day 113 and Day 365
GMC of anti-STm OAg, anti-SEn OAg and anti-Vi IgG before each study intervention administration [for infants 6 WOA] | At Day 1, Day 57 and Day 232
GMC of anti-STm OAg, anti-SEn OAg and anti-Vi IgG 28 days after each study intervention administration [for infants 6 WOA] | At Day 29, Day 85 and Day 260
Number of participants achieving at least 2-fold and 4fold increase in antiserotype specific IgG concentrations [for infants 6 MOA] | At 28 days after each study intervention administration (Day 29, Day 113 and Day 365) compared with before the first study intervention administration (Day 1)
Number of participants with anti-Vi IgG concentrations greater than or equal to (>=)2.0 micrograms per milliliter (µg/mL) and >=4.3 µg/mL [for infants 6 MOA] | Before each study intervention administration (Day 1, Day 85 and Day 337) and 28 days after each study intervention administration (Day 29, Day 113 and Day 365)
Number of participants achieving at least 2-fold and 4fold increase in antiserotype specific IgG concentrations [for infants 6 WOA] | At 28 days after each study intervention administration (Day 29, Day 85 and Day 260), compared with before the first study intervention administration (Day 1)
Number of participants with anti-Vi IgG concentrations >=2.0 µg/mL and >=4.3 µg/mL [for infants 6 WOA] | Before each study intervention administration (Day 1, Day 57 and Day 232) and 28 days after each study intervention administration (Day 29, Day 85 and Day 260)

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf